CLINICAL TRIAL: NCT01004081
Title: Phase 2a, Open-Label, Randomized, Noncomparative Study of BIIB021 in Combination With Exemestane in Women With Hormone Receptor-Positive, Advanced Metastatic Breast Cancer Who Have Progressed on a Nonsteroidal Aromatase Inhibitor
Brief Title: Hormone Receptor Positive Metastatic Breast Cancer (HR+ mBC) BIIB021 Plus Aromasin Schedule Finding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120BC201
Record Dates: First submitted 2009-09-18; First posted 2009-10-29 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
Keywords: Cancer of Breast; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — 6-chloro-9-(4-methoxy-3,5-dimethylpyridin-2-ylmethyl)-9H-purin-2-ylamine; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIIB021 BID + exemestane (Experimental): BIIB021 100 mg BID + exemestane 25 mg QD
  Interventions: Drug: BIIB021; Drug: exemestane (Aromasin)
- BIIB021 TIW + exemestane (Experimental): BIIB021 450 mg TIW + exemestane 25 mg QD
  Interventions: Drug: BIIB021; Drug: exemestane (Aromasin)

INTERVENTIONS:
Drug: BIIB021 — BID orally for 28 days
  Other Names: CNF2024
  Arms: BIIB021 BID + exemestane
Drug: BIIB021 — TIW orally for 28 days
  Other Names: CNF2024
  Arms: BIIB021 TIW + exemestane
Drug: exemestane (Aromasin) — Daily in tablet form for 28 days
  Other Names: Aromasin

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of 2 dosing regimens of BIIB021 in combination with exemestane in women whose HR+ breast cancer had progressed following treatment with a nonsteroidal aromatase inhibitor (AI).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age
* Must have histologically or cytologically confirmed estrogen receptor- positive or progesterone receptor-positive, incurable, locally advanced, or metastatic breast cancer.
* Must have disease progression during treatment with a nonsteroidal AI for locally advanced or metastatic disease, or relapse during treatment or within 12 months of discontinuation of treatment in the adjuvant setting.
* Must be a postmenopausal female.
* Must have measurable or evaluable disease.

  * Measurable disease is defined as >=1 lesion with a diameter of >=10 mm
  * Evaluable disease is defined as bone lesions evaluable by plain X ray, CT scan, or MRI. Lesions identified only by radionuclide bone scan are not allowed.
* One prior chemotherapy regimen for advanced mBC is allowed.
* Prior radiotherapy is allowed.
* Must be able to swallow and retain oral medication.
* ECOG performance status of <=2
* Required laboratory values

  * Plasma cortisol and adrenocorticotropic hormone (ACTH) levels that are not suggestive of adrenal insufficiency unless on replacement therapy for known adrenal insufficiency.

Exclusion Criteria:

* HER2 overexpressing tumor.
* History of central nervous system (CNS) metastasis.
* Previous treatment with exemestane or treatment with an Hsp90 inhibitor.
* Use of proton pump inhibitors.
* Known history of or positive test result for hepatitis B or C or HIV.
* History of gastrectomy or major surgery to small intestine.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the efficacy of 2 dosing regimens of BIIB021 in combination with exemestane in women whose HR+ breast cancer had progressed following treatment with a nonsteroidal AI. | As specified in protocol

SECONDARY OUTCOMES:
The secondary objective of this study is to evaluate the safety and tolerability of BIIB021 in combination with exemestane in this study population. | As specified in protocol

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (33):
- United States (18):
  - Research Site, Alabaster, Alabama
  - Research Site, Encinitas, California
  - Research Site, Gilroy, California
  - Research Site, Long Beach, California
  - Research Site, Davie, Florida
  - Research Site, Orlando, Florida
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Berkeley Heights, New Jersey
  - Research Site, New York, New York
  - Research Site, Fargo, North Dakota
  - Research Site, Columbus, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Lacey, Washington
- Australia (6):
  - Research Site, Waratah, New South Wales
  - Research Site, Wollongong, New South Wales
  - Research Site, Herston, Queensland
  - Research Site, Redcliffe, Queensland
  - Research Site, Hobart, Tasmania
  - Research Site, Geelong, Victoria
- Belgium (5):
  - Research Site, Brasschaat
  - Research Site, Edegem
  - Research Site, Kortrijk
  - Research Site, Liège
  - Research Site, Mons
- Russia (4):
  - Research Site, Kuzmolovskiy
  - Research Site, Moscow
  - Research Site, Ryazan
  - Research Site, Saint Petersburg